CLINICAL TRIAL: NCT00908154
Title: Single-blind, Randomised, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Repeat Doses of GSK1014802 and Its Interaction With Food in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Repeat Doses of GSK1014802.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 107727; SCB107727
Record Dates: First submitted 2009-05-07; First posted 2009-05-25 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Bipolar Depression; Bipolar Disorder
Keywords: sodium channel blocker; bipolar disorder; repeat dose
MeSH Terms: conditions — Bipolar Disorder | interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Cohort 1 (Other)
  Interventions: Drug: Placebo; Drug: GSK1014802
- Cohort 4 (Other)
  Interventions: Drug: Placebo; Drug: GSK1014802
- Cohort 3 (Other)
  Interventions: Drug: Placebo; Drug: GSK1014802
- Cohort 2 (Other)
  Interventions: Drug: Placebo; Drug: GSK1014802

INTERVENTIONS:
Drug: Placebo — Tablets to match GSK1014802
Drug: GSK1014802 — Sodium channel blocker
  Other Names: BIIB074 and CNV1014802

SUMMARY:
GSK1014802 is a use-dependent sodium channel blocker and an effective anticonvulsant in animal models.

This study is being conducted to obtain information regarding the safety, tolerability and pharmacokinetics of repeated doses of GSK1014802 administered for up to 28 days in healthy male or female subjects. In addition, the effect of food on the pharmacokinetics of GSK1014802 will be investigated.

DETAILED DESCRIPTION:
This study, previously posted by GlaxoSmithKline (GSK), was transitioned to Convergence Pharmaceuticals, Ltd., which spun off from GSK. Convergence Pharmaceuticals, Ltd., has now been acquired by Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.

  * Male or female (of non-child bearing potential) subjects aged between 18 and 55 years.
  * A female subject is eligible to participate if she is of non-childbearing potential.
  * Male subjects must agree to use an acceptable form of contraception.
  * Body weight ≥ 50 kg and BMI within the range 19 - 29.9 kg/m2 (inclusive)
  * Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
  * QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen.

  * A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
  * A positive test for HIV antibody.
  * History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females).
  * Current or past history of symptomatic orthostatic hypotension or history of unexplained vasovagal episode(s).
  * The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives (60 h) or twice the duration of the biological effect of the investigational product (whichever is longer).
  * Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
  * Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
  * History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
  * Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
  * Pregnant females.
  * Lactating females.
  * Unwillingness or inability to follow the procedures outlined in the protocol.
  * History of sensitivity to heparin or heparin-induced thrombocytopenia.
  * Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
  * . Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
  * History of known or suspected seizures, including infantile febrile, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05-31 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2008-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated by monitoring AEs and concomitant medication, ECG, Lead II monitoring, Holter monitoring, vital signs, and laboratory parameters. | 14-28 days
Blood concentrations of GSK1014802 following a single oral dose of GSK1014802. | 1 day
Blood concentrations of GSK1014802 following repeated oral doses of GSK1014802 given once daily or twice daily and their relationship with the GSK1014802 exposure after a single dose. | 14-28 days
Blood concentrations of GSK1014802 following repeated oral doses of GSK1014802 given once daily with or without food. | 14-28 days

SECONDARY OUTCOMES:
Bond-Lader VAS scale | 14-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Medical Director, Study Director — Biogen
Locations (1):
- GSK Investigational Site, London, United Kingdom